CLINICAL TRIAL: NCT05684731
Title: A Single-Arm, Open-Label Clinical Study to Evaluate the Safety, Tolerance and Preliminary Efficacy of KM1 Oncolytic Vaccinia Virus Injection Combined With Chemotherapy in Subjects With Recurrent or Refractory Ovarian Cancer
Brief Title: Safety and Efficacy of KM1 in Subjects With Recurrent or Refractory Ovarian Cancer
Acronym: K19017-004
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); People's Hospital of Quzhou (Other); Shenzhen Hua Yao Kang Ming Biopharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-TJ-KM1
Record Dates: First submitted 2023-01-03; First posted 2023-01-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
Keywords: KM1; oncolytic virus; immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: The study is a multicenter, open label, non-controlled, exploratory study. The "3+3" dose escalation design will be implemented to evaluate the safety and tolerability of KM1 in the treatment of subjects with recurrent or refractory ovarian cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: KM1 + Chemotherapy (Experimental): Biological: KM1 Administer via intraperitoneal infusion for 3 or 6 doses Q3D.
  Drug: Chemotherapy: Physician's Choice of carboplatin (preferred) or cisplatin，gemcitabine, taxane (paclitaxel, docetaxel or nab-paclitaxel) or pegylated liposomal doxorubicin，with or without bevacizumab.
  Administer beginning in Week 5 or Week 6.
  Interventions: Biological: KM1; Drug: Chemotherapy

INTERVENTIONS:
Biological: KM1 — Administer via intraperitoneal infusion for 3 or 6 doses Q3D.
Drug: Chemotherapy — Physician's Choice of carboplatin (preferred) or cisplatin，gemcitabine, taxane (paclitaxel, docetaxel or nab-paclitaxel) or pegylated liposomal doxorubicin，with or without bevacizumab.
  Administer beginning in Week 5 or Week 6.

SUMMARY:
The purpose of this study is to determine if KM1 is well tolerated with anti-tumor activity in patients diagnosed with recurrent or refractory ovarian cancer, and explore the Recommend Phase 2 Dose (RP2D) of KM1 in the treatment of patients with recurrent or refractory ovarian cancer.

DETAILED DESCRIPTION:
Oncolytic virus therapy is a kind of immunotherapy that can selectively infect and kill tumor cells without damaging normal cells. It has shown good therapeutic effects in the treatment of various types of tumors. KM1 is a genetically modified recombinant vaccinia virus, which has good therapeutic effect on many solid tumors, including ovarian cancer. This study includes Phase Ia and Phase Ib. In the Phase Ia study, subjects will receive three doses intraperitoneal infusion of KM1 followed by chemotherapy. In the Phase Ib study, subjects will receive six doses intraperitoneal infusion of KM1 preceding chemotherapy. Subjects will be followed in the study for 6 months after last dose of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytopathology confirmed epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer, except mucinous cancer.
* Relapsed/refractory subjects who failed to receive systemic treatment (at least one standard platinum containing regimen); Note: If the disease relapses, there should be evidence showing imaging or clinical progress (such as cytological report of new ascites or pleural effusion). Only the increase of CA125 cannot be used as the standard of disease recurrence.
* Performance status ECOG of 0 or 1.
* Life expectancy of at least 3 months.
* Toxicities of prior therapies have not been resolved to Grade 1 or baseline (except for alopecia, pigmentation or other toxicity considered as no safety risk to the subject in the study).
* At least 1 measurable target lesion by RECIST 1.1.
* Adequate renal, hepatic, bone marrow function, adequate coagulation tests, adequate immune function by lymphocyte count.
* Pregnancy test results within 14 days before the treatment were negative. Subjects of childbearing age must agree to use at least one medically approved contraceptive measure (such as surgical sterilization, oral contraceptives, intrauterine devices, sexual desire control, etc.) during the study treatment and at least 6 months after the last trial drug treatment;
* Subjects voluntarily participated in the study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* • Central nervous system (CNS) metastasis or cancerous meningitis (Note: Subjects with treated CNS metastases may participate in this trial if the subject is neurologically stable ≥3 months).

  * Prior malignancy of other histology active within previous 3 years except for locally curable cancers apparently cured such as basal/squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of cervix or breast.
  * Received any of the following treatments within a specific time frame prior to enrollment:

    1. Have received surgery of Grade II or above within 4 weeks (Whether or not related to tumor), except minimally invasive surgery under gastrointestinal endoscopy;
    2. Have received radiotherapy within 2 weeks (the investigator can judge the appropriate time of enrollment according to the patient's toxicity recovery after radiotherapy);
    3. Within 4 weeks or participating in other therapeutic/interventional clinical studies;
    4. Have received local anti-tumor treatment within 4 weeks;
  * Allergic to the test drug or its active ingredients and excipients.
  * Has had severe allergic reaction after receiving smallpox vaccine in the past.
  * Has a history of severe skin diseases requiring systemic treatment within 2 years, such as eczema, atopic dermatitis, burns, seborrheic dermatitis, psoriasis, severe acne, etc.
  * Has had an allogenic tissue/solid organ transplant.
  * Active infection or fever of unknown cause (>38.5 ℃).
  * Active pulmonary tuberculosis (TB) who are receiving anti tuberculosis treatment or who have received anti tuberculosis treatment within 1 year before screening;
  * Positive anti-HIV (+) or anti-HCV (+) or syphilis specific antibody (TPHA) or active hepatitis B.
  * Has a history of serious cardiovascular or cerebrovascular diseases, including but not limited to:

    1. New York Heart Association (NYHA) congestive heart failure of grade III or above;
    2. Serious arrhythmia requiring drug treatment;
    3. Acute myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass grafting, and stenting occurred within 6 months;
    4. Left ventricular ejection fraction (EF)<60%;
    5. QTcF interval ≥ 460 ms, or there are risk factors of torsade de pointes ventricular tachycardia, such as hypokalemia, family history of long QT syndrome or family history of arrhythmia (such as preexcitation syndrome);
    6. Presence of uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic BP>100 mmHg).
  * Active autoimmune diseases such as inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autohemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis), but the following conditions are allowed to enter the screening: type I diabetes, hypothyroidism that can be controlled only through alternative treatment, skin diseases that do not need systemic treatment (such as vitiligo, psoriasis or alopecia).
  * Symptomatic malignant ascites or pleural effusions defined as rapidly progressive ascites with abdominal distension and gastrointestinal dysfunction, pleural effusions with respiratory difficulties requiring frequent paracentesis > once every 14 days.
  * Contraindications for intraperitoneal (IP) catheter placement: Bowel obstruction with distended abdomen, rigid abdomen with bulky anterior wall carcinomatosis, abdominal wall hernia mesh that precludes laparoscopic entry to abdomen.
  * Active gastrointestinal bleeding.
  * Accompanied by unstable mental illness, alcohol abuse, drug abuse or drug abuse.
  * Other conditions that investigator considers unsuitable for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | From baseline during treatment to 21 days following last dose of KM1.
  Type and incidence of dose-limiting toxicity (DLT) by dose group
Adverse events (AEs) and serious adverse events (SAEs) | From baseline during treatment to 21 days following last dose of KM1
  Type and incidence of adverse events (AEs) and serious adverse events (SAEs) by dose group
Maximum tolerable dose (MTD)/ Recommended Phase II Dose (RP2D） | From baseline during treatment to 21 days following last dose of KM1.

SECONDARY OUTCOMES:
Virus particles | From baseline during treatment to 21 days following last dose of KM1.
  Level of virus particles tested by plaque assay in blood, body fluids (urine, feces and saliva), peritoneal fluid (if any), and tumor tissue (if any) at baseline and during treatment period.
Virus coding genes | From baseline during treatment to 21 days following last dose of KM1.
  Level of virus coding genes tested by PCR assay in blood, body fluids (urine, feces and saliva), peritoneal fluid (if any), and tumor tissue (if any) at baseline and during treatment period.
Anti-Drug Antibodies (ADA) | From baseline during treatment to 21 days following last dose of KM1.
  Titer of positive ADA against KM1 at baseline and during treatment period.
Progression Free Survival (PFS) by RECIST 1.1 | From date of randomization up to 6 months following last dose of chemotherapy.
  Time from study treatment initiation to the first occurrence of disease progression or death (of any cause).
Objective Response Rate (ORR) by RECIST 1.1 | From date of randomization up to 6 months following last dose of chemotherapy.
  The ratio of the sum of Complete Response & Partial Response divided by the number of participants from the start of treatment to confirmation of response.
Disease Control Rate (DCR) RECIST 1.1 | From date of randomization up to 6 months following last dose of chemotherapy.
  The ratio of the sum of Complete Response & Partial Response & Stable Disease divided by the number of participants from the start of treatment to confirmation of response
CA-125 Response | From date of randomization up to 6 months following last dose of chemotherapy.
  Level of CA-125 (UI/ml) at baseline and after treatment measured by Enzyme Linked Immunosorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD. PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No